CLINICAL TRIAL: NCT05076331
Title: Health and Aging Brain Study: Health Disparities Tau PET Scan Study
Brief Title: Health and Aging Brain Study: Health Disparities Tau Positron Emission Tomography (PET) Scan Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of North Texas Health Science Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-125
Record Dates: First submitted 2021-09-28; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; Tau PET Scan; Health Disparities; Brain Aging
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health and Aging Brain Study Cohort: Health and Aging Brain Study participants age 50 and older.
  Interventions: Diagnostic Test: PI-2620 tracer for Tau PET scan

INTERVENTIONS:
Diagnostic Test: PI-2620 tracer for Tau PET scan — Tau PET scans are obtained using PI-2620 tracer provided by Life Medical Imaging.

SUMMARY:
The purpose of this project is to study the aging brain among participants enrolled in the Health and Aging Brain Study: Health Disparities project . There are a number of things that can influence how people think as they age, including diabetes, depression, as well as our biology. In this study, the investigators seek to study the aging brain by using brain PET scans that create detailed pictures of the brain.

DETAILED DESCRIPTION:
There are a number of things that can influence how we think as people age, including diabetes, depression, as well as our biology. In this study, the investigators are using PET scans with a tracer to create detailed pictures of the brain. This information will be used to help the investigators understand how the brain ages and in the future could be used to develop better diagnostics and treatments for Alzheimer's disease and memory loss in Mexican Americans, African Americans, and non-Hispanic whites. The goal of this study is to address this disparity by enrolling ethnically diverse participants in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in the Health and Aging Brain Study HD: Health Disparities project
2. Provided consent to re-contact
3. Willing and capable of undergoing PET scan of the head

Exclusion Criteria:

1. Inability to provide informed consent by self or by proxy.
2. Pregnant or breast feeding women*
3. History of alcoholism or drug dependency/abuse within the last 2 years before screening
4. Hypersensitivity to the active substance or to any of the following excipients is contraindicated: sodium dihydrogen phosphate, phosphoric acid, sodium ascorbate, ethanol (anhydrous), water for injection
5. Participants may not be in this study if they do not meet the safety criteria to undergo imaging procedures.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants of the multi ethnic "Health and Aging Brain Study Health Disparities" .Men and women age 50 and above that may or may not have cognitive impairment. .
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Health Disparities in Aging | Through study completion in 2 years
  Examine the prevalence of Tau burden among a multi ethnic cohort

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Texas Health Science Center, Fort Worth, Texas, United States